CLINICAL TRIAL: NCT05319314
Title: A Phase 1 Multicenter Study Evaluating the Safety and Tolerability of GCC19CART for Subjects With Relapsed or Refractory Metastatic Colorectal Cancer
Brief Title: GCC19CART for Patients With Metastatic Colorectal Cancer
Acronym: CARAPIA-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Cellular Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICT-GCC19CART-US-001
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: relapsed metastatic colorectal cancer; refractory metastatic colorectal cancer; chimeric antigen receptors (CAR); colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GCC19CART (Experimental): Single infusion of GCC19CART at the dose assigned to an individual subject.
  All subjects will receive the same investigational therapy with the dose administered dependent upon the dose level they are assigned to in a sequential manner.
  Two dose level escalations are planned with one dose de-escalation listed if needed.
  Interventions: Drug: GCC19CART

INTERVENTIONS:
Drug: GCC19CART — Single infusion of Chimeric Antigen Receptor (CAR) transduced autologous T cells administered intravenously (i.v.)

SUMMARY:
Study ICT-GCC19CART-US-001 (CARAPIA-1) is a Phase 1 study evaluating the safety, tolerability, clinical activity, pharmacokinetics and pharmacodynamics of GCC19CART in subjects with relapsed or refractory metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Clinical and histopathological diagnosis of metastatic colorectal cancer
* Guanylate Cyclase (GCC) positive disease as determined by immunohistochemistry (IHC). Positivity on staining of archival tumor tissue is adequate.
* Limited liver disease (less than 7 lesions with largest lesion less than 3 cm)
* No surgical options with curative intent.
* Received prior therapy with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy in the advanced or metastatic setting, an anti-vascular endothelial growth factor (anti-VEGF) biological therapy if not contraindicated, and if RAS wild-type an anti-epidermal growth factor receptor (anti-EGFR) therapy in a manner consistent with National Comprehensive Cancer Network (NCCN) guidelines. Treatment must have been discontinued for disease progression or intolerance to therapy.
* Have at least one extracranial measurable target lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 standard.

Exclusion Criteria:

* Subjects with tumor lesion(s) in a location that may cause perforation of an organ or structure (such as the digestive track, urinary bladder, or blood vessel) with GCC19CART therapy.
* No active infectious diseases or comorbid conditions that would interfere with safety or data quality.
* Subjects with active infection requiring systemic therapy or causing fever (temperature > 38.1˚C) or subjects with unexplained fever (temperature > 38.1˚C) within 7 days prior to enrollment (leukapheresis) and reconfirmed prior to the day of investigational product administration.
* Pregnant or breast-feeding women

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) defined as dose-limiting toxicities (DLTs) during 3+3 dose escalation study | Infusion (Day 0) up to Day 28
Maximum tolerable dose (MTD) based on incidence of dose-limiting toxicities (DLTs) during 3+3 dose escalation study | Infusion (Day 0) up to Day 28
Recommended Phase 2 dose (RP2D) based on incidence of dose-limiting toxicities (DLTs) during 3+3 dose escalation study | Infusion (Day 0) up to Day 28

SECONDARY OUTCOMES:
Best overall response as measured by overall response rate based on the tumor size per Response Evaluation Criteria in Solid Tumors RECIST Version 1.1 | Infusion (Day 0) up to approximately 12 months or until disease progression/recurrence
Duration of Response (DOR) | Infusion (Day 0) up to approximately 12 months
  The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Progression Free Survival (PFS) | Day 30 (date of leukapheresis) up to approximately 13 months or until the earliest date of disease progression per RECIST 1.1, or death from any cause, whichever comes first.
  Progression free survival (PFS) time which is defined as time from date of leukapheresis until the earliest date of disease progression per RECIST 1.1, or death from any cause, whichever comes first.
Overall Survival (OS) | Day 30 (date of leukapheresis) up to approximately 13 months or until death from any cause
  Overall survival (OS) is defined as the time from the date of leukapheresis until death from any cause.
Copy number of Guanylate Cyclase C (GCC) by Quantitative Polymerase Chain Reaction (qPCR) | Infusion, Inpatient Monitoring and Post Treatment Period (Up to 12 months)
Copy number of each individual CD19 by Quantitative Polymerase Chain Reaction (qPCR) | Infusion, Inpatient Monitoring and Post Treatment Period (Up to 12 months)
Cytokine level in serum | Infusion (Day 0) up to 12 months post treatment
AUC0 - Tmax: The area under curve (AUC) from time zero to Tmax in peripheral blood (days x copies/μg) | Infusion (Day 0) up to 12 months post treatment
AUCTmax - 28d and/or AUCTmax - 84d: The area under curve (AUC) from time Tmax to day 28 and/or AUCTmax - 84d or other disease assessment days, in peripheral blood (days x copies/μg) | Infusion (Day 0) up to 12 months post treatment
AUC0 - 28d and/or AUC0 - 84d: The area under curve (AUC) from time zero to day 28 and/or day 84 in peripheral blood (days x copies/μg) | Infusion (Day 0) up to 12 months post treatment
Cmax: The maximum (peak) observed in peripheral blood or other body fluid drug concentration after single dose administration (copies/μg) | Infusion (Day 0) up to 12 months post treatment
Tmax: The time to reach maximum(peak) in peripheral blood or other body fluid drug concentration after single dose administration (days) | Infusion (Day 0) up to 12 months post treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Baylor Scott & White Research Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No